CLINICAL TRIAL: NCT01334684
Title: White Blood Cells Gene Expression Profiles as a Tool for Predicting Metformin Efficacy in Patients With Type 2 Diabetes Mellitus
Brief Title: Gene Expression Profiles and Metformin Efficacy in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: University Hospital, Catania (Other)
Responsible Party: Salvatore De Cosmo, Casa Sollievo della Sofferenza IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GExpProMet
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Metformin Efficacy; Gene Expression Profiles; Personalized Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Other): At study entry, all oral hypoglycemic agents will be discontinued for 5 days and then metformin (2,550 mg/daily) will be given for 3 months. Fasting plasma glucose will be measured at baseline and 3 months after metformin treatment. Patients will be stratified according to the median value of metformin efficacy as indicated by fasting glucose change after metformin treatment (i.e. baseline fasting glucose minus 3-month fasting glucose).
  So, two subgroups of patients will be obtained, defined as relatively "high responders" (individual fasting glucose change > median value) or relatively "low responders" (individual fasting glucose change < median value) to metformin monotherapy.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin, pills, 850 mg three times a day for three months

SUMMARY:
Our general aim is to investigate whether messenger RNA (mRNA) and/or microRNA (miRNA) expression profiles in white blood cells, predict metformin monotherapy efficacy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (duration of diabetes of at least 2 years)
* age 40-70 yrs
* HbA1c > 6.4 < 9.0

Exclusion Criteria:

* insulin therapy
* contraindications to metformin use

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose change after metformin treatment in respect to mRNA and miRNA expression profiles in white blood cells | Baseline and after three months of metfomin therapy
  Changes in fasting glucose levels will be used to evaluate if metformin monotherapy efficacy in type 2 diabetic patients is predicted by mRNA and/or miRNA expression profiles.
  Please note that metformin major effect is to decrease hepatic glucose output and, therefore, to lower fasting plasma glucose which is, in fact, the clinical outcome used in this study.
  Finally, because of a very short wash-out period (i.e. 5 days) we will not be able to use HbA1c which will be inevitably conditioned by previous oral hypoglicemic therapy.

SECONDARY OUTCOMES:
Change in fasting insulin levels after metformin treatment in respect to mRNA and miRNA expression profiles in white blood cells | Baseline and after three months of metfomin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore De Cosmo, MD, Study Chair — Casa Sollievo della Sofferenza IRCCS
Locations (1):
- Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Foggia, Italy

REFERENCES:
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Iwao-Koizumi K, Matoba R, Ueno N, Kim SJ, Ando A, Miyoshi Y, Maeda E, Noguchi S, Kato K. Prediction of docetaxel response in human breast cancer by gene expression profiling. J Clin Oncol. 2005 Jan 20;23(3):422-31. doi: 10.1200/JCO.2005.09.078. PMID 15659489
- [Background] Bertucci F, Finetti P, Rougemont J, Charafe-Jauffret E, Nasser V, Loriod B, Camerlo J, Tagett R, Tarpin C, Houvenaeghel G, Nguyen C, Maraninchi D, Jacquemier J, Houlgatte R, Birnbaum D, Viens P. Gene expression profiling for molecular characterization of inflammatory breast cancer and prediction of response to chemotherapy. Cancer Res. 2004 Dec 1;64(23):8558-65. doi: 10.1158/0008-5472.CAN-04-2696. PMID 15574762
- [Background] Ayers M, Symmans WF, Stec J, Damokosh AI, Clark E, Hess K, Lecocke M, Metivier J, Booser D, Ibrahim N, Valero V, Royce M, Arun B, Whitman G, Ross J, Sneige N, Hortobagyi GN, Pusztai L. Gene expression profiles predict complete pathologic response to neoadjuvant paclitaxel and fluorouracil, doxorubicin, and cyclophosphamide chemotherapy in breast cancer. J Clin Oncol. 2004 Jun 15;22(12):2284-93. doi: 10.1200/JCO.2004.05.166. Epub 2004 May 10. PMID 15136595
- [Background] Xia L, Zhang D, Du R, Pan Y, Zhao L, Sun S, Hong L, Liu J, Fan D. miR-15b and miR-16 modulate multidrug resistance by targeting BCL2 in human gastric cancer cells. Int J Cancer. 2008 Jul 15;123(2):372-379. doi: 10.1002/ijc.23501. PMID 18449891
- [Background] Blower PE, Chung JH, Verducci JS, Lin S, Park JK, Dai Z, Liu CG, Schmittgen TD, Reinhold WC, Croce CM, Weinstein JN, Sadee W. MicroRNAs modulate the chemosensitivity of tumor cells. Mol Cancer Ther. 2008 Jan;7(1):1-9. doi: 10.1158/1535-7163.MCT-07-0573. Epub 2008 Jan 9. PMID 18187804
- [Background] Sarasin-Filipowicz M, Krol J, Markiewicz I, Heim MH, Filipowicz W. Decreased levels of microRNA miR-122 in individuals with hepatitis C responding poorly to interferon therapy. Nat Med. 2009 Jan;15(1):31-3. doi: 10.1038/nm.1902. Epub 2009 Jan 4. PMID 19122656
- [Background] Wingrove JA, Daniels SE, Sehnert AJ, Tingley W, Elashoff MR, Rosenberg S, Buellesfeld L, Grube E, Newby LK, Ginsburg GS, Kraus WE. Correlation of peripheral-blood gene expression with the extent of coronary artery stenosis. Circ Cardiovasc Genet. 2008 Oct;1(1):31-8. doi: 10.1161/CIRCGENETICS.108.782730. PMID 20031539
- [Background] Rosenberg S, Elashoff MR, Beineke P, Daniels SE, Wingrove JA, Tingley WG, Sager PT, Sehnert AJ, Yau M, Kraus WE, Newby LK, Schwartz RS, Voros S, Ellis SG, Tahirkheli N, Waksman R, McPherson J, Lansky A, Winn ME, Schork NJ, Topol EJ; PREDICT (Personalized Risk Evaluation and Diagnosis in the Coronary Tree) Investigators. Multicenter validation of the diagnostic accuracy of a blood-based gene expression test for assessing obstructive coronary artery disease in nondiabetic patients. Ann Intern Med. 2010 Oct 5;153(7):425-34. doi: 10.7326/0003-4819-153-7-201010050-00005. PMID 20921541
- [Background] Yakeu G, Butcher L, Isa S, Webb R, Roberts AW, Thomas AW, Backx K, James PE, Morris K. Low-intensity exercise enhances expression of markers of alternative activation in circulating leukocytes: roles of PPARgamma and Th2 cytokines. Atherosclerosis. 2010 Oct;212(2):668-73. doi: 10.1016/j.atherosclerosis.2010.07.002. Epub 2010 Jul 16. PMID 20723894
- [Background] Camargo A, Ruano J, Fernandez JM, Parnell LD, Jimenez A, Santos-Gonzalez M, Marin C, Perez-Martinez P, Uceda M, Lopez-Miranda J, Perez-Jimenez F. Gene expression changes in mononuclear cells in patients with metabolic syndrome after acute intake of phenol-rich virgin olive oil. BMC Genomics. 2010 Apr 20;11:253. doi: 10.1186/1471-2164-11-253. PMID 20406432